CLINICAL TRIAL: NCT02015195
Title: Efficacy of Topical Agents in the Treatment of Chrysaora Chinensis Stings
Brief Title: Effective Treatments for Jellyfish Stings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul S Auerbach, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JSP-001
Record Dates: First submitted 2013-12-04; First posted 2013-12-19 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Jellyfish Stings
Keywords: Jellyfish stings; Treatment; Humans; Topical Treatments; Pain; Erythema
MeSH Terms: conditions — Pain; Erythema | interventions — Acetic Acid; Ammonia; Lidocaine; 2-Propanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Acetic Acid 5% (Experimental): Acetic Acid (5%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Interventions: Other: Acetic Acid (5%); Other: No treatment
- Sodium Bicarbonate Slurry (50%) (Experimental): Sodium Bicarbonate Slurry (50%) Dosage form: Liquid slurry Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Interventions: Other: Sodium Bicarbonate Slurry (50%); Other: No treatment
- Papain Slurry (70%) (Experimental): Papain Slurry (70%) Dosage form: Liquid slurry Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Interventions: Other: Papain Slurry (70%); Other: No treatment
- Household ammonia (10%) (Experimental): Ammonia (10%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Interventions: Other: Ammonia (10%); Other: No treatment
- Lidocaine (4%) (Experimental): Lidocaine (4%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Interventions: Drug: Lidocaine (4%); Other: No treatment
- Isopropyl Alcohol (70%) (Experimental): Isopropyl Alcohol (70%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Interventions: Other: Isopropyl Alcohol (70%); Other: No treatment
- Hot Water (40 degrees Celsius) (Experimental): Hot Tap Water (40 degrees Celsius) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Interventions: Other: Hot Tap Water (40 degrees Celsius); Other: No treatment

INTERVENTIONS:
Other: Acetic Acid (5%)
  Other Names: Vinegar
  Arms: Acetic Acid 5%
Other: Sodium Bicarbonate Slurry (50%)
  Arms: Sodium Bicarbonate Slurry (50%)
Other: Papain Slurry (70%)
  Other Names: Adolfo's Meat tenderizer
  Arms: Papain Slurry (70%)
Other: Ammonia (10%)
  Other Names: Household ammonia
  Arms: Household ammonia (10%)
Drug: Lidocaine (4%)
  Other Names: Liquid Lidocaine
  Arms: Lidocaine (4%)
Other: Isopropyl Alcohol (70%)
  Other Names: Rubbing alcohol
  Arms: Isopropyl Alcohol (70%)
Other: Hot Tap Water (40 degrees Celsius)
  Other Names: Hot Water
  Arms: Hot Water (40 degrees Celsius)
Other: No treatment
  Other Names: Nothing is given topically to treat sting. This is the control.

SUMMARY:
The purpose of the study is to attempt to determine which treatment from commonly used treatments is the best at reducing pain and redness of the skin after a sting from a Portuguese Man of War, Chrysaora chinensis, or Chrysaora fuscescens.

Jellyfish stings are a common occurrence in many parts of the world causing significant morbidity to persons stung by jellyfish while participating in marine activities whether commercial or recreational. Much debate and confusion exist both in the medical literature and the common recommendations regarding how to treat persons stung by jellyfish. Specifically concerning what topical treatments are most efficacious at decreasing envenomation by nematocyst on skin, preventing the firing of un-discharged nematocyst, decreasing inflammation and pain resulting from envenomation by nematocyst. Antidotal recommendations and past studies have referenced numerous different topical treatments for jellyfish stings including but not limited to vinegar, urine, alcohol, distilled spirits, ammonia, bleach, acetone, bicarbonate slurry, lidocaine, meat tenderizer, Coca Cola, old wine, salt water, cold packs, hot water, and commercial products such as Stingose and Stingaid. Conflicting data exists regarding what works and what does not for nematocysts discharge, skin erythema, and pain reaction.

The investigators would like to investigate which treatment is best out of some of the more commonly studied treatments for reducing pain and erythema.

The investigators would like to complete a research study to try to bring some reasonable evidence to the field treatment of jellyfish stings, namely, the decontamination process (e.g., what can you put on a jellyfish sting that will be helpful, based on real data?).

The questions asked are as follows:

* What topical treatments for jellyfish stings actually decrease the amount of inflammation seen on a macroscopic level on the skin of humans?
* What topical treatments for jellyfish stings actually decrease the sensation of pain in humans?
* Do topical chemical treatments cause different outcomes when exposed to the above parameters?
* Do different species of jellyfish nematocysts react differently based on the type of topical chemical treatment used? What is the variation of effects of topical treatments based on the species of jellyfish sting?

Specifically, the investigators will be stinging human subject on both arms with a segment of tentacle for approximately 2 minutes. This will be followed by no treatment on one arm (control arm) and by treatment on the other arm with either: acetic acid (5%), sodium bicarbonate slurry (50%), papain slurry (70%), ammonia (10%), viscous lidocaine (4%), isopropyl alcohol (70%), or hot tap water (40 degrees Celsius). Outcomes measured will include pain and erythema.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* Healthy volunteers

Exclusion Criteria:

* Known history of allergic reaction or anaphylaxis to prior Cnidaria sting of there envenomations
* Family history of anaphylaxis to any sting from either Cnidaria, bee, or wasp
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Auerbach, MD, Principal Investigator — Division of Emergency Medicine, Stanford University Medical Center; Matthieu P DeClerck, MD, Study Director — Division of Emergency Medicine, Stanford University Hospital
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy human subjects were recruited by advertisement on Stanford University campus during the months of May and June, 2013 for a study that took place within a medical ward within a hospital during July, 2013. 97 patients were enrolled.
Pre-assignment Details: Volunteers were excluded if they were pregnant, had a history of allergic reaction to prior jellyfish or insect sting, a family history of severe allergic reaction to jellyfish or insect sting, or a history of heart or lung disease.
Groups:
- Acetic Acid 5%: Acetic Acid (5%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Acetic Acid (5%)
  No treatment
  The left arm was always the active treatment arm; the right arm was the "control" arm (i.e., no treatment).
- Sodium Bicarbonate Slurry (50%): Sodium Bicarbonate Slurry (50%) Dosage form: Liquid slurry Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Sodium Bicarbonate Slurry (50%)
  No treatment
  The left arm was always the active treatment arm; the right arm was the "control" arm (i.e., no treatment).
- Papain Slurry (70%): Papain Slurry (70%) Dosage form: Liquid slurry Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Papain Slurry (70%)
  No treatment
  The left arm was always the active treatment arm; the right arm was the "control" arm (i.e., no treatment).
- Household Ammonia (10%): Ammonia (10%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Ammonia (10%)
  No treatment
  The left arm was always the active treatment arm; the right arm was the "control" arm (i.e., no treatment).
- Lidocaine (4%): Lidocaine (4%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Lidocaine (4%)
  No treatment
  The left arm was always the active treatment arm; the right arm was the "control" arm (i.e., no treatment).
- Isopropyl Alcohol (70%): Isopropyl Alcohol (70%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Isopropyl Alcohol (70%)
  The left arm was always the active treatment arm; the right arm was the "control" arm (i.e., no treatment).
  No treatment
- Hot Water (40 Degrees Celsius): Hot Tap Water (40 degrees Celsius) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Hot Tap Water (40 degrees Celsius)
  No treatment
  The left arm was always the active treatment arm; the right arm was the "control" arm (i.e., no treatment).
Period: Overall Study
Arm/Group | Acetic Acid 5% | Sodium Bicarbonate Slurry (50%) | Papain Slurry (70%) | Household Ammonia (10%) | Lidocaine (4%) | Isopropyl Alcohol (70%) | Hot Water (40 Degrees Celsius)
Started | 16 | 16 | 16 | 1 | 16 | 16 | 16
Completed | 16 | 16 | 16 | 0 | 16 | 16 | 16
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: one patient treated with ammonia - adverse local skin reaction - this treatment arm therefore withdrawn from study
Groups:
- Acetic Acid 5%: Acetic Acid (5%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Acetic Acid (5%)
  No treatment
  11 males, 5 females treated
- Sodium Bicarbonate Slurry (50%): Sodium Bicarbonate Slurry (50%) Dosage form: Liquid slurry Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Sodium Bicarbonate Slurry (50%)
  No treatment
  8 males, 8 females treated
- Papain Slurry (70%): Papain Slurry (70%) Dosage form: Liquid slurry Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Papain Slurry (70%)
  No treatment
  9 males, 7 females treated
- Household Ammonia (10%): Ammonia (10%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Ammonia (10%)
  No treatment
  1 female treated; adverse local skin reaction; study arm therefore withdrawn
- Lidocaine (4%): Lidocaine (4%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Lidocaine (4%)
  No treatment
  10 males, 6 females treated
- Isopropyl Alcohol (70%): Isopropyl Alcohol (70%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Isopropyl Alcohol (70%)
  No treatment
  8 makes, 8 females treated
- Heated Water (40 Degrees Celsius): Hot Tap Water (40 degrees Celsius) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Heated Tap Water (40 degrees Celsius)
  No treatment
  8 males, 8 females treated
- Total: Total of all reporting groups
Arm/Group | Acetic Acid 5% | Sodium Bicarbonate Slurry (50%) | Papain Slurry (70%) | Household Ammonia (10%) | Lidocaine (4%) | Isopropyl Alcohol (70%) | Heated Water (40 Degrees Celsius) | Total
Number analyzed (Participants) | 16 | 16 | 16 | 1 | 16 | 16 | 16 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 16 | 1 | 16 | 16 | 16 | 97
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 7 | 1 | 6 | 8 | 8 | 43
  Male | 11 | 8 | 9 | 0 | 10 | 8 | 8 | 54
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 16 | 1 | 16 | 16 | 16 | 97

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Pain in the Treated Human Arm (Not Placebo) From Baseline Determined by Measures (17) Taken Over 24 Hours
Description: Pain is measured on a scale of 1-10 with 0 being no pain and 10 being worse pain ever felt. Baseline pain will be measured immediately after being stung for 2 minutes without any treatment. Subsequent pain felt at every 2 minutes for 30 minutes, at 1 hour post sting, and at 24 hours post sting will be based on changes from the original baseline pain. Mean change is defined as the mean change in pain from all time points measured from each participant and then averaged for each group. The control arm (placebo) was collected and analyzed in parallel to the treatment arm. The "mean change" for the treatment arm was then compared with the "mean change" for the control arm as a baseline. Hence, the data presented are the estimated effect for each treatment group compared to the control arms for each group.
Time Frame: 24 hours
Population: one participant excluded because of adverse local skin reaction to household ammonia
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Acetic Acid 5%: Acetic Acid (5%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Acetic Acid (5%)
  No treatment
- Sodium Bicarbonate Slurry (50%): Sodium Bicarbonate Slurry (50%) Dosage form: Liquid slurry Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Sodium Bicarbonate Slurry (50%)
  No treatment
- Papain Slurry (70%): Papain Slurry (70%) Dosage form: Liquid slurry Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Papain Slurry (70%)
  No treatment
- Lidocaine (4%): Lidocaine (4%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Lidocaine (4%)
  No treatment
- Isopropyl Alcohol (70%): Isopropyl Alcohol (70%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Isopropyl Alcohol (70%)
  No treatment
- Hot Water (40 Degrees Celsius): Hot Tap Water (40 degrees Celsius) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Hot Tap Water (40 degrees Celsius)
  No treatment
Arm/Group | Acetic Acid 5% | Sodium Bicarbonate Slurry (50%) | Papain Slurry (70%) | Lidocaine (4%) | Isopropyl Alcohol (70%) | Hot Water (40 Degrees Celsius)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
units on a scale | 0.13 [-0.31 to 0.55] | -0.19 [-0.63 to 0.25] | -0.46 [-0.90 to -0.01] | -0.31 [-0.76 to 0.126] | -0.26 [-0.70 to 0.17] | 0.42 [-0.02 to 0.87]

2. Primary Outcome: Mean Change in Erythema (Redness) in the Treated Human Arm (Not Placebo) From Baseline Determined by Measures (3) Taken Over 24 Hours
Description: Visual inspection of sting sites will be done at 30 minutes post sting (after treatment completed), 1 hour post sting, and 24 hours post sting. Erythema Index (EI) imeasures increase in cutaneous vasodilation. A computer-measured (Image-J software) EI was used to remove subjectivity. A numeric score was created for the level of erythema, with "0" representing baseline erythema on the control arm. Any positive number indicates more and negative number less erythema on treatment arm compared to placebo. EI values were measured on a "scale" from -20 to +20 with "0" being the midpoint where there would be equal amounts of erythema on both the treatment and control arm. The erythema they experienced on the "treatment arm" was then measured as more erythema (a positive value up to 20) or less erythema (a negative value up to -20).
Time Frame: 30 minutes, 1 hour, and 24 hours
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Acetic Acid 5% | Sodium Bicarbonate Slurry (50%) | Papain Slurry (70%) | Lidocaine (4%) | Isopropyl Alcohol (70%) | Hot Water (40 Degrees Celsius)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
units on a scale | 4.43 [-3.52 to 12.39] | -12.07 [-19.26 to -4.88] | 0.58 [-7.37 to 8.55] | -4.14 [-11.56 to 3.27] | 2.11 [-5.84 to 10.07] | -4.11 [-11.79 to 3.56]

ADVERSE EVENTS:
Groups:
- Household Ammonia (10%): Ammonia (10%) Dosage form: Liquid Dosage: 5 ml topical Frequency: every 2 minutes Duration: 30 minutes
  Ammonia (10%)
  No treatment
  The first patient treated had an adverse local skin reaction, so this study arm was discontinued
Arm/Group | Acetic Acid 5% | Sodium Bicarbonate Slurry (50%) | Papain Slurry (70%) | Household Ammonia (10%) | Lidocaine (4%) | Isopropyl Alcohol (70%) | Hot Water (40 Degrees Celsius)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/1 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 1/1 | 0/16 | 0/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetic Acid 5% (N=16) | Sodium Bicarbonate Slurry (50%) (N=16) | Papain Slurry (70%) (N=16) | Household Ammonia (10%) (N=1) | Lidocaine (4%) (N=16) | Isopropyl Alcohol (70%) (N=16) | Hot Water (40 Degrees Celsius) (N=16)
erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — erythema
pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No